CLINICAL TRIAL: NCT00894972
Title: Examining the Effectiveness of a Post-operative Rehabilitation Program Emphasizing Restoration of Multifidus Muscle Function for Individuals Undergoing Lumbar Discectomy: a Randomized Clinical Trial
Brief Title: Rehabilitation Following Lumbar Disc Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Julie Fritz, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32474
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Lumbar Disc Herniation; Radiculopathy
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy | interventions — Diskectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): General exercise. Participants in this group will perform aerobic exercise, range of motion exercise and general strengthening exercise.
  Interventions: Other: Rehabilitation following lumbar disc surgery (discectomy)
- 2 (Experimental): Specific exercise. Participants in this group will perform aerobic exercise, range of motion exercise, and specific motor control exercises.
  Interventions: Other: Rehabilitation following lumbar disc surgery (discectomy)

INTERVENTIONS:
Other: Rehabilitation following lumbar disc surgery (discectomy) — Exercise: walking, range of motion, and general trunk strengthening with or without specific trunk muscle motor control exercises.

SUMMARY:
The proposed study will be a randomized clinical trial designed to determine the most effective physical therapy program for individuals who have undergone lumbar discectomy surgery. The study will compare two different post-operative physical therapy programs (general strengthening or general + specific strengthening). Both groups will begin treatment 2 weeks post-surgery. Subjects in both groups will receive weekly treatment sessions for 8 weeks with a treatment program emphasizing exercises shown to activate the large trunk muscles without imposing potentially harmful compression or shear forces. The general + specific strengthening group will also receive exercises shown to isolate activation of the deep trunk muscles, in particular the multifidus, with training augmented by the use of diagnostic ultrasound biofeedback. Patient assessments will be conducted pre- and post-surgery, as well as 10 (post-treatment) and 26 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Diagnosis of LDH based on imaging (MRI or CT scan) of the lumbar spine with concurring clinical examination findings (based on the judgment of the attending neurosurgeon)
* Appropriate surgical candidate based on the opinion of the attending spine surgeon, and scheduled for single-level lumbar discectomy (open or micro-discectomy).
* Able to attend weekly treatment sessions.

Exclusion Criteria:

* Prior surgery to the lumbar spine
* Spondylolytic or degenerative spondylolisthesis present on pre-surgical imaging
* Unable to speak and understand English
* Peri- or post-operative complication (infection, nerve injury, dural tear, vascular injury, etc.) that would limit or delay the ability to participate in post-operative rehabilitation.
* Multi-level surgery or the use of instrumentation during surgery (i.e., lumbar fusion)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry disability index | Preoperative, 2 postoperative weeks, 10 postoperative weeks, 6 postoperative months

SECONDARY OUTCOMES:
Lumbar multifidus muscle activation as estimated by diagnostic ultrasound imaging | preoperative, 2 postoperative weeks, 10 postoperative weeks, 6 postoperative months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fritz, PT, PhD, ATC, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Department of Physical Therapy, Salt Lake City, Utah, United States